CLINICAL TRIAL: NCT03086473
Title: A Randomized, Placebo-controlled Trial of Early Caffeine in Preterm Neonates
Brief Title: Early Caffeine in Preterm Neonates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jennifer Shepherd (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor-Investigator, Jennifer Shepherd, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HS-15-00899
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: BPD - Bronchopulmonary Dysplasia; Apnea of Prematurity; Hemodynamic Instability; Intubation
Keywords: caffeine; intubation; hemodynamics; mechanical ventilation; cardiac output; near infrared spectroscopy; functional echocardiography
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Apnea | interventions — caffeine citrate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Each participant is assigned to one of two arms of the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant and participant's parents, medical care providers, and investigators will remain masked to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Caffeine (Other): Participant will receive caffeine citrate 20mg/kg IV within 2 hours of life and placebo (normal saline IV) at 12 hours of life. Both infusions will be of identical volumes and appearance, and will be administered over 30 minutes.
  Interventions: Drug: Caffeine Citrate
- Placebo (Other): Participant will receive placebo (normal saline IV) within 2 hours of life and caffeine citrate 20mg/kg IV at 12 hours of life. Both infusions will be of identical volumes and appearance, and will be administered over 30 minutes.
  Interventions: Drug: Placebo (Normal Saline)

INTERVENTIONS:
Drug: Caffeine Citrate — The intervention in this study is timing of the initial caffeine dose. In the Caffeine arm, participants will receive Caffeine Citrate 20mg/kg IV (volume dose 1ml/kg) within 2 hours of life, and Normal Saline (0.9% NaCl) 1ml/kg IV at 12 hours of life.
  Other Names: Cafcit
  Arms: Caffeine
Drug: Placebo (Normal Saline) — The intervention in this study is timing of the initial caffeine dose. In the Placebo arm, participants will receive Normal Saline (0.9%NaCl) 1ml/kg IV within 2 hours of life, and Caffeine Citrate 20mg/kg IV (volume dose 1ml/kg) at 12 hours of life.
  Arms: Placebo

SUMMARY:
This is a clinical trial which will investigate whether administration of caffeine, a respiratory stimulant, to preterm babies soon after birth can prevent the need for a breathing tube, or intubation. Many preterm babies who require intubation are intubated soon after birth, often within the first few hours. If caffeine is given early enough and is sufficient to stimulate effective breathing, perhaps these babies may not require intubation. Additionally, caffeine may improve blood flow in preterm babies when given soon after birth. Approximately half of babies in this study will receive caffeine within two hours after birth, and half will receive caffeine 12 hours after birth. The hypothesis is that preterm babies who receive caffeine within 2 hours after birth will have a lower incidence of intubation than preterm babies who receive caffeine 12 hours after birth. The main secondary hypothesis is that caffeine given soon after birth will enhance blood flow in preterm babies.

DETAILED DESCRIPTION:
Caffeine is routinely administered to extremely preterm neonates as a respiratory stimulant to prevent or treat apnea of prematurity, or prolonged pauses in breathing in preterm babies. Caffeine, a methylxanthine, is an adenosine receptor antagonist that has the effects of relaxing smooth muscle in the airways, stimulating the central nervous system and cardiac muscle, and acting as a diuretic. The mode of action in apnea of prematurity could be from several mechanisms, including stimulation of respiratory drive, enhancement of minute ventilation, increased response to hypercapnia, increase in skeletal muscle tone, and decrease in diaphragmatic fatigue.

The timing of caffeine administration is highly variable, ranging from the first hours of life to several days after birth. In the Caffeine for Apnea of Prematurity (CAP) trial, in which the average day of initial caffeine dose was 3 days of life, the incidence of bronchopulmonary dysplasia (BPD) was significantly reduced in the caffeine group compared to the placebo group (47% vs 36%, p<0.001). Neonates in the caffeine group also had fewer days of mechanical ventilation and oxygen exposure, both of which are known risk factors in the development of BPD. Further studies have demonstrated greater benefit of caffeine given in the first 2-3 days of life versus later. These studies suggest that caffeine administered earlier in life may be beneficial in terms of respiratory outcomes. However, the effects of caffeine administered shortly after birth are unknown and need to be studied with a randomized, placebo-controlled trial.

The investigators postulate that by giving caffeine as soon as possible after birth, intrinsic respiratory function will be supported sufficiently to avoid intubation altogether, thus eliminating a major risk factor for BPD. Intravenous caffeine reaches therapeutic level almost immediately, typically within thirty minutes of administration. However, the majority of infants who require invasive ventilation are intubated within the first few hours of life, usually before the infant has received caffeine. Additionally, many centers utilize minimally invasive administration of surfactant, a medication that helps keep lungs open by lowering surface tension, to treat respiratory distress syndrome of the newborn in attempt to avoid intubation, as preterm neonates who do not require immediate intubation and instead receive non-invasive continuous positive airway pressure (CPAP) at birth have decreased risk of BPD. These techniques require spontaneous, effective breathing, and early caffeine administration may aid in this process. This study aims to deliver caffeine to preterm infants immediately after birth to determine whether intubation can be avoided.

While the primary outcome of this study is aimed at reducing intubation rates and thus affecting rates of BPD, beneficial cardiovascular effects may also be noted. The incidence of hypotension in preterm infants <28 weeks is as high as 78%.This study will also be using non-invasive technologies to continuously monitor hemodynamic parameters including cardiac function, output, blood flow, oxygenation to the brain surrounding the administration of caffeine. Very early caffeine therapy may improve cardiovascular function in this early transitional period, potentially decreasing the risk of devastating complications of prematurity such as intraventricular hemorrhage.

This is a double-blinded, randomized, placebo-controlled clinical trial which will investigate whether administration of caffeine to preterm neonates (<32 weeks' gestation) within the first 2 hours of life compared to 12 hours of life will decrease the rate of intubation during the first 12 hours of life. This study will also investigate whether caffeine administration to preterm neonates (<32 weeks' gestation) increases cardiac output. A total of 88 infants will be included in this study, randomized to two study arms. One arm will receive intravenous caffeine citrate within 2 hours of life and placebo (normal saline) at 12 hours of life, and the other arm will receive placebo within 2 hours of life and caffeine citrate at 12 hours of life. Therefore, all participants will receive caffeine by 12 hours of life, and the only variable is the timing of caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Neonates <32 weeks' gestational age born at LAC+USC Medical Center, Hollywood Presbyterian Medical Center, or other sites affiliated with USC or CHLA will be considered for enrollment.

Exclusion Criteria:

* Exclusions are major congenital anomalies, major cardiac defects (other than patent ductus arteriosus, patent foramen ovale, small atrial septal defect, and small ventricular septal defect), and intubation in the delivery room
* If intravenous access is not obtained within the first 2 hours of life (either through peripheral IV or central venous catheter), then the neonate will no longer be eligible for the study.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Intubation | Within 12 hours of life
  Need for endotracheal intubation within the first 12 hours of life.

SECONDARY OUTCOMES:
Cardiac output | Prior to and 1 hour after receipt of caffeine/placebo at 2 hours of life and 12 hours of life
  Changes in cardiac output after administration of caffeine.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Shepherd, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Hollywood Presbyterian Medical Center, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Northway WH Jr, Rosan RC, Porter DY. Pulmonary disease following respirator therapy of hyaline-membrane disease. Bronchopulmonary dysplasia. N Engl J Med. 1967 Feb 16;276(7):357-68. doi: 10.1056/NEJM196702162760701. No abstract available. PMID 5334613
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Long-term effects of caffeine therapy for apnea of prematurity. N Engl J Med. 2007 Nov 8;357(19):1893-902. doi: 10.1056/NEJMoa073679. PMID 17989382
- [Background] Lodha A, Seshia M, McMillan DD, Barrington K, Yang J, Lee SK, Shah PS; Canadian Neonatal Network. Association of early caffeine administration and neonatal outcomes in very preterm neonates. JAMA Pediatr. 2015 Jan;169(1):33-8. doi: 10.1001/jamapediatrics.2014.2223. PMID 25402629
- [Background] Logan JW, O'Shea TM, Allred EN, Laughon MM, Bose CL, Dammann O, Batton DG, Engelke SC, Leviton A; ELGAN Study Investigators. Early postnatal hypotension and developmental delay at 24 months of age among extremely low gestational age newborns. Arch Dis Child Fetal Neonatal Ed. 2011 Sep;96(5):F321-8. doi: 10.1136/adc.2010.183335. Epub 2010 Dec 7. PMID 21138828
- [Background] Laptook AR, O'Shea TM, Shankaran S, Bhaskar B; NICHD Neonatal Network. Adverse neurodevelopmental outcomes among extremely low birth weight infants with a normal head ultrasound: prevalence and antecedents. Pediatrics. 2005 Mar;115(3):673-80. doi: 10.1542/peds.2004-0667. PMID 15741371
- [Background] Aranda JV, Beharry K, Valencia GB, Natarajan G, Davis J. Caffeine impact on neonatal morbidities. J Matern Fetal Neonatal Med. 2010 Oct;23 Suppl 3:20-3. doi: 10.3109/14767058.2010.517704. PMID 20873976
- [Background] Patel RM, Leong T, Carlton DP, Vyas-Read S. Early caffeine therapy and clinical outcomes in extremely preterm infants. J Perinatol. 2013 Feb;33(2):134-40. doi: 10.1038/jp.2012.52. Epub 2012 Apr 26. PMID 22538326
- [Background] Dobson NR, Patel RM, Smith PB, Kuehn DR, Clark J, Vyas-Read S, Herring A, Laughon MM, Carlton D, Hunt CE. Trends in caffeine use and association between clinical outcomes and timing of therapy in very low birth weight infants. J Pediatr. 2014 May;164(5):992-998.e3. doi: 10.1016/j.jpeds.2013.12.025. Epub 2014 Jan 23. PMID 24461786
- [Background] Aranda JV, Cook CE, Gorman W, Collinge JM, Loughnan PM, Outerbridge EW, Aldridge A, Neims AH. Pharmacokinetic profile of caffeine in the premature newborn infant with apnea. J Pediatr. 1979 Apr;94(4):663-8. doi: 10.1016/s0022-3476(79)80047-5. PMID 430317
- [Background] More K, Sakhuja P, Shah PS. Minimally invasive surfactant administration in preterm infants: a meta-narrative review. JAMA Pediatr. 2014 Oct;168(10):901-8. doi: 10.1001/jamapediatrics.2014.1148. PMID 25089718
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Background] Cunningham S, Symon AG, Elton RA, Zhu C, McIntosh N. Intra-arterial blood pressure reference ranges, death and morbidity in very low birthweight infants during the first seven days of life. Early Hum Dev. 1999 Dec;56(2-3):151-65. doi: 10.1016/s0378-3782(99)00038-9. PMID 10636594
- [Background] Cordero L, Timan CJ, Waters HH, Sachs LA. Mean arterial pressures during the first 24 hours of life in < or = 600-gram birth weight infants. J Perinatol. 2002 Jul-Aug;22(5):348-53. doi: 10.1038/sj.jp.7210736. PMID 12082467
- [Background] Kluckow M, Evans N. Low superior vena cava flow and intraventricular haemorrhage in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F188-94. doi: 10.1136/fn.82.3.f188. PMID 10794784
- [Background] Sheth RD. Trends in incidence and severity of intraventricular hemorrhage. J Child Neurol. 1998 Jun;13(6):261-4. doi: 10.1177/088307389801300604. PMID 9660508
- [Background] Noori S, McCoy M, Anderson MP, Ramji F, Seri I. Changes in cardiac function and cerebral blood flow in relation to peri/intraventricular hemorrhage in extremely preterm infants. J Pediatr. 2014 Feb;164(2):264-70.e1-3. doi: 10.1016/j.jpeds.2013.09.045. Epub 2013 Oct 30. PMID 24183212
- [Background] Soloveychik V, Bin-Nun A, Ionchev A, Sriram S, Meadow W. Acute hemodynamic effects of caffeine administration in premature infants. J Perinatol. 2009 Mar;29(3):205-8. doi: 10.1038/jp.2008.193. Epub 2008 Dec 4. PMID 19052555
- [Background] Walther FJ, Erickson R, Sims ME. Cardiovascular effects of caffeine therapy in preterm infants. Am J Dis Child. 1990 Oct;144(10):1164-6. doi: 10.1001/archpedi.1990.02150340110035. PMID 2403102
- [Background] Hoecker C, Nelle M, Poeschl J, Beedgen B, Linderkamp O. Caffeine impairs cerebral and intestinal blood flow velocity in preterm infants. Pediatrics. 2002 May;109(5):784-7. doi: 10.1542/peds.109.5.784. PMID 11986437
- [Background] Tracy MB, Klimek J, Hinder M, Ponnampalam G, Tracy SK. Does caffeine impair cerebral oxygenation and blood flow velocity in preterm infants? Acta Paediatr. 2010 Sep;99(9):1319-23. doi: 10.1111/j.1651-2227.2010.01828.x. PMID 20412101
- [Background] Soleymani S, Borzage M, Noori S, Seri I. Neonatal hemodynamics: monitoring, data acquisition and analysis. Expert Rev Med Devices. 2012 Sep;9(5):501-11. doi: 10.1586/erd.12.32. PMID 23116077
- [Background] Noori S, Wlodaver A, Gottipati V, McCoy M, Schultz D, Escobedo M. Transitional changes in cardiac and cerebral hemodynamics in term neonates at birth. J Pediatr. 2012 Jun;160(6):943-8. doi: 10.1016/j.jpeds.2011.12.008. Epub 2012 Jan 11. PMID 22244465
- [Background] Noori S, Drabu B, Soleymani S, Seri I. Continuous non-invasive cardiac output measurements in the neonate by electrical velocimetry: a comparison with echocardiography. Arch Dis Child Fetal Neonatal Ed. 2012 Sep;97(5):F340-3. doi: 10.1136/fetalneonatal-2011-301090. PMID 22933092
- [Background] Noori S, Anderson M, Soleymani S, Seri I. Effect of carbon dioxide on cerebral blood flow velocity in preterm infants during postnatal transition. Acta Paediatr. 2014 Aug;103(8):e334-9. doi: 10.1111/apa.12646. Epub 2014 Apr 29. PMID 24673183
- [Background] Ma M, Noori S, Maarek JM, Holschneider DP, Rubinstein EH, Seri I. Prone positioning decreases cardiac output and increases systemic vascular resistance in neonates. J Perinatol. 2015 Jun;35(6):424-7. doi: 10.1038/jp.2014.230. Epub 2015 Jan 15. PMID 25590219
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Katheria AC, Sauberan JB, Akotia D, Rich W, Durham J, Finer NN. A Pilot Randomized Controlled Trial of Early versus Routine Caffeine in Extremely Premature Infants. Am J Perinatol. 2015 Jul;32(9):879-86. doi: 10.1055/s-0034-1543981. Epub 2015 Jan 21. PMID 25607226